CLINICAL TRIAL: NCT04467996
Title: Evaluation of the Minimum Effective Duration of Intrauterine Balloon Tamponade for the Management of Postpartum Hemorrhage: A Randomized Controlled Trial
Brief Title: Minimum Effective Duration of Intrauterine Balloon Tamponade for the Management of Postpartum Hemorrhage
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Denver Health and Hospital Authority (Other)
Responsible Party: Principal Investigator, LARREANICOLE, Obstetrician Gynegologist, Assistant Professor, Denver Health and Hospital Authority
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 19-3070
Record Dates: First submitted 2020-07-08; First posted 2020-07-13 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Postpartum Hemorrhage, Immediate
MeSH Terms: conditions — Postpartum Hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- 6 hour IUBT placement (Active Comparator)
  Interventions: Device: Intrauterine balloon tamponade
- 18 hour IUBT placement (Active Comparator)
  Interventions: Device: Intrauterine balloon tamponade

INTERVENTIONS:
Device: Intrauterine balloon tamponade — Intrauterine balloon will be placed in the uterus for postpartum hemorrhage control.

SUMMARY:
Intrauterine balloon tamponade (IUBT) is recommended worldwide as the second-line therapy to treat postpartum hemorrhage. While much literature demonstrates the effectiveness of this therapy, little is known about how long the IUBT should be used once placed. Though it is common to use IUBT for 12-24 hours, the balloon may be equally effective when used for shorter durations of time, which could have beneficial effects for patients and hospitals. The proposed study is a pragmatic randomized controlled trial of non-inferiority comparing two durations of time for intrauterine balloon tamponade placement, 6 and 18 hours, in controlling postpartum hemorrhage.

The specific aims of the proposed study are to determine: 1) whether quantitative blood loss significantly differs when the balloon is removed in 6 hours compared to 18 hours, 2) whether hemorrhage-related morbidity differs when the IUBT is kept in place for 6 or 18 hours, and 3) whether shorter duration of IUBT placement has beneficial effects including shortened postpartum hospital stays, improved maternal-infant bonding, and reduced postpartum pain prior to maternal discharge from hospital.

We hypothesize that, once hemorrhage control has been achieved with IUBT placement, there is no clinically significant difference in postpartum blood loss when the balloon is removed 6 hours after placement compared to 18 hours after placement.

ELIGIBILITY:
Inclusion Criteria:

* Women at Denver Health and Hospital Authority (DHHA) who have an IUBT placed for postpartum hemorrhage due to uterine atony will be approached for enrollment in the study.

Exclusion Criteria:

* Women will be excluded from the study if they: are less than 18 years of age; had a cesarean delivery; are unable to consent for themselves; have a preexisting or acquired clotting factor disorder such as von Willebrand or hemophilia, disseminated intravascular coagulation, or therapeutic anticoagulation at time of delivery; would refuse blood product transfusion; have a fetal demise or birth of a previable fetus; or are incarcerated at the time of delivery. Women who do not speak English or Spanish will be offered enrollment if a phone interpreter is available to review the consent, but will be excluded from the survey portion of the study.

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 64 (Estimated)
Dates: Start 2020-10-19 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Quantitative blood loss | 18 hours
  total blood loss includes output from the intrauterine balloon plus blood loss from sanitary pads

SECONDARY OUTCOMES:
Postpartum hemorrhage related outcomes | during admission
  return to the OR, replacement of the IUBT, hysterectomy, pelvic artery embolization
Hematocrit | during admission
  change in hematocrit from admission to discharge
Postpartum length of stay | during admission
  Length of stay in hours
Endometritis | during admission
  diagnosed postpartum
Chorioamnionitis | during admission
  requiring more than one dose of antibiotics postpartum
Transfusion of packed red blood cells | during admission
  after IUBT placement
Maternal-infant bonding | during admission
  measured by the mother-to-infant bonding scale (MIBS), scale 0-27, higher score indicates worse maternal-infant bonding
Maternal pain | during admission
  measured by the visual analogue scale (VAS), scale 0-10, higher score indicates worse pain

CONTACTS AND LOCATIONS:
Locations (1):
- Denver Health Hospital, Denver, Colorado, United States

IPD SHARING:
Plan to Share IPD: Undecided